CLINICAL TRIAL: NCT02877771
Title: Tandem Predictive Low Glucose Suspend Inpatient Feasibility Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 010300
Record Dates: First submitted 2016-08-09; First posted 2016-08-24 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes; Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

ARMS (1):
- t:slim insulin pump with predictive low glucose suspend (Experimental): To assess the functionality of a predictive low glucose suspend (PLGS) system that uses CGM values to suspend basal insulin delivery when hypoglycemia is predicted as well as resume basal insulin delivery once Continuous Glucose Monitoring (CGM) values begin to increase.
  Interventions: Device: t:slim insulin pump with predictive low glucose suspend

INTERVENTIONS:
Device: t:slim insulin pump with predictive low glucose suspend — To assess the functionality of a predictive low glucose suspend (PLGS) system that uses Continuous Glucose Monitoring (CGM) values to suspend basal insulin delivery when hypoglycemia is predicted as well as resume basal insulin delivery once Continuous Glucose Monitoring (CGM) values begin to increase.

SUMMARY:
The goal of this study is to assess the functionality of an integrated predictive low glucose suspend system designed to minimize the incidence and duration of hypoglycemia by suspending insulin delivery if hypoglycemia is projected.

DETAILED DESCRIPTION:
This protocol is designed to test the functionality of a predictive low glucose suspend system under supervised conditions where basal insulin rates are manually increased until a system generated suspension occurs. The study will collect data that will be used for planning a pivotal study, and the study data are intended to be used to support a Premarket Approval (PMA) application.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes requiring insulin therapy for at least 12 months
* Insulin pump therapy for at least 6 months
* Age ≥18.0 years
* Subject demonstrates stable insulin regimen including basal rates, insulin sensitivity factor and insulin:carbohydrate ratio for at least 3 months

Exclusion Criteria:

* Pregnant (female subjects must have negative urine or serum pregnancy screening test)
* Severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrollment
* Diabetic ketoacidosis in the month prior to enrollment
* A current condition that would prevent the use of a CGM sensor or insulin pump, or in the judgment of the investigator is a contraindication to study participation
* Use of acetaminophen during study participation
* Current use of any medication intended to lower glucose other than insulin including naturaceuticals, oral or non-insulin injectable medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Suspension of Insulin Delivery | 8 hours between 9pm and 5am
  To test functionality of the system
Restoration of insulin delivery | 8 hours between 9pm and 5am
  To test functionality of the system
Agreement between algorithm-recommended pump action | 8 hours between 9pm and 5am
  To test functionality of the system

OTHER OUTCOMES:
Duration of insulin suspension | 8 hours between 9pm and 5am
  To test functionality of the system
Continuous Glucose Monitoring (CGM) glucose nadir | 8 hours between 9pm and 5am
  To test functionality of the system
Reference blood glucose | 8 hours between 9pm and 5am
  To test functionality of the system

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado